CLINICAL TRIAL: NCT03747653
Title: A Phase I, Multicentre, Open-label, Self-control Study to Evaluate the Pharmacokinetics of Recombinant Human Coagulation Factor VIII-Fc Fusion Protein for Injection in Adolescent and Adult Patients With Hemophilia A
Brief Title: A Study to Evaluate the Pharmacokinetics of Recombinant Human Coagulation Factor VIII-Fc Fusion Protein for Injection
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Kaifeng Pharmaceutical (Group) Co., Ltd. (Industry)
Collaborators: Beijing Furen Biomedical Research Institute Co., Ltd. (Unknown)
Responsible Party: Sponsor
Other Study IDs: CTR20182090
Record Dates: First submitted 2018-11-12; First posted 2018-11-20 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Hemophilia A
Keywords: Hemophilia A; Pharmacokinetics; Factor VIII-Fc Fusion Protein; Adolescent and Adult Patients; Phase I; Safety and Tolerability
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm 1: Participants will receive a single intravenous (i.v.) injection of ADVATE followed by a single intravenous (i.v.) injection of Recombinant Human Coagulation Factor VIII-Fc fusion protein for Injection (FRSW107) at a low dose.
  Interventions: Drug: ADVATE; Drug: FRSW107
- Arm 2: Participants will receive a single intravenous (i.v.) injection of ADVATE followed by a single intravenous (i.v.) injection of Recombinant Human Coagulation Factor VIII-Fc fusion protein for Injection (FRSW107) at a high dose.
  Interventions: Drug: ADVATE; Drug: FRSW107

INTERVENTIONS:
Drug: ADVATE — Patients will be administered a single dose of ADVATE.
Drug: FRSW107 — Patients will be administered a single dose of FRSW107 for Injection.

SUMMARY:
Primary objective: To assess the pharmacokinetics of Recombinant Human Coagulation Factor VIII-Fc fusion protein for Injection at two dose levels in patients with hemophilia A.

Secondary objectives: To assess Safety and Tolerability by monitoring FVIII recovery and adverse events in patients with hemophilia A.

ELIGIBILITY:
Inclusion Criteria:

* 12 years to 60 years, male.
* The activity of the coagulation factor VIII (FVIII:C) < 2%, and previously treated with FVIII concentrate (s) for a minimum of 150 exposure days (EDs) prior to study entry.
* Non-immune deficiency (CD4 > 200/μL).
* Non-acute hemorrhagic state.
* No history of a positive inhibitor test (< 0.6 BU) or clinical signs of decreased response to FVIII administrations. No Family history of inhibitors.
* Platelet count > 100,000 platelets/μL.
* Normal prothrombin time or INR < 1.3.
* Normal thrombin time (TT).
* Normal previous results of vWF antigen examination.
* Negative lupus anticoagulant .
* Capable of understanding and willing to comply with the conditions of the protocol have read (patient and/or guardian).

Exclusion Criteria:

* Hypersensitive to any of the excipients of the test materials (e.g. allergic to murine or hamster origin heterologous proteins).
* History of hypersensitivity or anaphylaxis associated with any FVIII or IgG2 administration.
* Current FVIII inhibitor-positive or history of FVIII inhibitor-positive.
* Other coagulation disorder(s) in addition to hemophilia A.
* Infusion of any products containing FVIII within 4 days prior screening or within 72 h prior to administration.
* Patients with severe heart disease, including myocardial infarction, heart failure (III or higher level).
* Clinically significant of other systematic diseases: alcoholism, drug abuse, mental disorders and mental retardation.
* Significant hepatic or renal impairment (ALT and AST > 2×ULN; serum bilirubin level > 3 × upper limit of normal (ULN) , BUN > 2×ULN, Cr > 2.0 mg/dL).
* One or more clinically significant tests for Human Immunodeficiency Virus (HIV), Antisyphilitic spirulina (TPHA) and Hepatitis C Virus (HCV) Antibody.
* Patients who received any anticoagulant or antiplatelet therapy within one week prior screening or need to receive an anticoagulant or antiplatelet therapy during the period of clinical trials.
* Patients having major surgery or receiving blood or bood components transfusion within 4 weeks prior screening or having planned major surgery schedule during the study.
* Patients who previously participated in the other clinical trials within 1 month prior screening.
* Any life-threatening disease or condition which, according to the investigator's judgment, could not benefit from the trial participation.
* Patient who is considered by the other investigators not suitable for clinical study.

Ages: 12 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Hemophilia A is an X-chromosome-linked recessive inherited bleeding disorder caused by a deficiency of coagulation factor VIII (FVIII).
Study Population: Adolescent and Adult patients with Hemophilia A from clinical registration.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2019-03-08 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Maximum measured concentration of FVIII:C (Cmax). | Pre-dose and post dose of FRSW107 up to 10 days.
  Measured by the One-stage aPTT Clotting Assay.
Time required for the concentration of the drug to reach half of its original value (T1/2). | Pre-dose and post dose of FRSW107 up to 10 days.
  Measured by the One-stage aPTT Clotting Assay.
Area Under the Curve to Infinity (AUC). | Pre-dose and post dose of FRSW107 up to 10 days.
  Measured by the One-stage aPTT Clotting Assay.
The measure of the efficiency of the body to remove the drug and the unit is the volume of the plasma or blood cleared of drug per unit time (CL). | Pre-dose and post dose of FRSW107 up to 10 days.
  Measured by the One-stage aPTT Clotting Assay.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE V5.0. | Post dose of FRSW107 up to 28.
  Adverse events related to Recombinant Human Coagulation Factor VIII-Fc fusion protein for Injection according to Common Terminology Criteria for Adverse Events (CTCAE) NCI.V5.0.
Development of Inhibitor. | Pre-dose and post dose of FRSW107 up to 28 days.
  Measured by the Nijmegen-Modified Bethesda Assay.

CONTACTS AND LOCATIONS:
Overall Officials: Renchi Yang, PhD, Principal Investigator — Institute of Hematology & Blood Diseases Hospital Chinese Academy of Medical Sciences & Peking Union Medical College
Locations (5):
- China (5):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Southern Medical University Nanfang Hospital, Guangzhou, Guangzhou
  - Jinan Central Hospital, Jinan, Shandong
  - Institute of Hematology & Blood Diseases Hospital Chinese Academy of Medical Sciences & Peking Union Medical College, Tianjin, Tianjin Municipality
  - Hematology Department, Beijing Children's Hospital, Capital Medical University, Beijing